CLINICAL TRIAL: NCT04594434
Title: Efficiency of the Use of Benevolent Memories in the EMDR Protocol in Complex Psychotrauma (Benevolence Study)
Brief Title: Eye Movement Desensitization and Reprocessing (EMDR) in Complex Psychotrauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A01914-35
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Complex Post-Traumatic Stress Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protocol EMDR + SB / SMP protocol (adjusted) (Experimental): Association of a positive memory with the "recommended" therapy based on EMDR.
  Interventions: Other: Scale SUD; Other: VOC scale; Other: DES II scale
- protocol EMDR (standard). (Active Comparator): "recommended" therapy based on EMDR.
  Interventions: Other: Scale SUD; Other: VOC scale; Other: DES II scale

INTERVENTIONS:
Other: Scale SUD — Subjective Units of Distress Scale ou Subjective Units of Disturbance Scale is a scale of subjective appreciation of emotions
Other: VOC scale — The VOC (Validity Of Cognition) scale is a scale of value given to cognition.
Other: DES II scale — The Dissociative Experiences Scale (DES), which is translated as the Dissociative Experiences Scale, is a self-questionnaire to assess the frequency of various dissociative symptoms in the patient's daily life.

SUMMARY:
This study wants to demonstrate the effectiveness of combining a positive memory with "recommended" therapy based on EMDR in reducing the disturbance that patients with complex psychotrauma may experience. The positive memory will be called "benevolent memory" (SB) or "less worse memory" (SMP).

DETAILED DESCRIPTION:
This is an interventional study, prospective, exploratory, comparative, randomized, controlled versus reference treatment protocol, open.

Patients will be seen 16 times for the purposes of the study. They will be hospitalized during therapy. Discharge from hospitalization occurs during follow-up depending on the patient's condition.

They will be evaluated over a period of 4 to 6 weeks between the start (Day 0 = Week 1) and the end of treatment (visit week 12). These visits will coincide with treatment sessions with the EMDR ± SB / SMP protocol, as part of the support of their complex psychotrauma. At the end of treatment, the patient will be evaluated during follow-up visits at Month 1, Month 3 and Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a combination of a period of complex trauma and a disturbance triggered by situations in adulthood;
* Having signed an informed consent form to participate in the study.

Exclusion Criteria:

* Protected patient (under legal protection, or deprived of liberty by judicial or administrative decision);
* Patient seeking legal benefit from participating in the study;
* Patient previously treated with EMDR;
* Patient unable to understand the information related to the study (linguistic, psychological, cognitive reason, etc.);
* Untreated epileptic patient;
* Patient with severe oculomotor disorders;
* Patient in hypomanic phase;
* Patient treated with high dose corticosteroids;
* Patient with alcohol and / or drug misuse in the 7 days preceding inclusion;
* Pregnant or likely to be (of childbearing age, without effective contraception) or breastfeeding;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not beneficiary of a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the combination of SB and / or PMS with EMDR technique on reducing the disturbance experienced by patients with complex psychotrauma. | 6 months
  Percentage of patients with a 50% reduction in the SUD score(44/5000 measured by the SUD scale ranging from 0 to 10) at the end of the 3rd "active" EMDR session compared to the pre-treatment score of the 1st "active" session

SECONDARY OUTCOMES:
Disturbance felt | 6 months
  The % of patients responding to therapy (with SUD scores = 0 and VOC = 7) at M1, M3 and M6 will be compared between the 2 groups by a Cochran-Mantel-Haenszel test.
Level of dissociation | 6 months
  The change in the level of dissociation by the DES II scale (score from 0 to 100) after therapy will be compared between the 2 groups by an analysis of covariance with adjustment for the score at inclusion;

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique d'Yveline, Vieille-Église-en-Yvelines, France